CLINICAL TRIAL: NCT04586010
Title: A Phase III Multicenter Randomized, Double-Blind, Double-Dummy, Parallel-Group Study to Evaluate the Efficacy and Safety of Fenebrutinib Compared With Teriflunomide in Adult Patients With Relapsing Multiple Sclerosis
Brief Title: A Study to Evaluate the Efficacy and Safety of Fenebrutinib Compared With Teriflunomide in Relapsing Multiple Sclerosis (RMS)
Acronym: FENhance
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GN41851; 2019-004857-10 (EudraCT Number); 2022-502609-14-00 (EU CTIS Number)
Record Dates: First submitted 2020-10-08; First posted 2020-10-14 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Relapsing Multiple Sclerosis
MeSH Terms: interventions — fenebrutinib; teriflunomide

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Sponsor will also be blinded.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Fenebrutinib (Experimental): Participants will receive oral fenebrutinib with teriflunomide-matching placebo.
  Interventions: Drug: Fenebrutinib; Drug: Placebo
- Teriflunomide (Active Comparator): Participants will receive oral teriflunomide with fenebrutinib-matching placebo in a blinded fashion.
  Interventions: Drug: Teriflunomide; Drug: Placebo

INTERVENTIONS:
Drug: Fenebrutinib — Participants will receive fenebrutinib.
  Arms: Fenebrutinib
Drug: Teriflunomide — Participants will receive teriflunomide.
  Arms: Teriflunomide
Drug: Placebo — Participants will receive teriflunomide-matching placebo or fenebrutinib-matching placebo.

SUMMARY:
A study to evaluate the efficacy and safety of fenebrutinib on disability progression and relapse rate in adult participants with RMS. Eligible participants will be randomized 1:1 to either fenebrutinib or teriflunomide. At the end of the DBT phase (after disclosure of the DBT results), the Sponsor will determine whether or not to initiate the open-label extension phase of the study.

ELIGIBILITY:
Inclusion Criteria:

* Expanded Disability Status Scale (EDSS) score of 0 - 5.5 at screening.
* A diagnosis of RMS in accordance with the revised 2017 McDonald Criteria.
* Ability to complete the 9-Hole Peg Test (9-HPT) for each hand in < 240 seconds.
* Ability to perform the Timed 25-Foot Walk Test (T25FWT) in <150 seconds.
* For female participants of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures, and refrain from donating eggs.
* For male participants: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures, and refrain from donating sperm.

OLE Inclusion Criteria:

* Completed the Double-Blind Treatment (DBT) phase of the study (remaining on study treatment; no other Disease-Modifying Therapy (DMT) administered) and who, in the opinion of the investigator, may benefit from treatment with fenebrutinib.
* Participants randomized to the teriflunomide treatment arm during the DBT phase must undergo the accelerated teriflunomide elimination procedure (ATEP) prior to the first administration of open-label fenebrutinib.
* For female participants of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures, and refrain from donating eggs.
* For male participants: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures, and refrain from donating sperm.

Exclusion Criteria:

* Disease duration of > 10 years from the onset of symptoms and an EDSS score at screening < 2.0.
* Female participants who are pregnant or breastfeeding, or intending to become pregnant.
* Male participants who intend to father a child during the study.
* A diagnosis of primary progressive MS (PPMS) or non-active secondary progressive MS (SPMS).
* Any known or suspected active infection at screening, including but not limited to a positive screening test for Hepatitis B and C, an active or latent or inadequately treated infection with tuberculosis (TB), a confirmed or suspected progressive multifocal leukoencephalopathy (PML).
* History of cancer including hematologic malignancy and solid tumors within 10 years of screening.
* Known presence of other neurological disorders, that could interfere with the diagnosis of MS or assessments of efficacy or safety during the study and clinically significant cardiovascular, psychiatric, pulmonary, renal, hepatic, endocrine, metabolic or gastrointestinal disease.
* Rare hereditary problems of galactose intolerance, total lactase deficiency, or glucose-galactose malabsorption.
* Hypoproteinemia.
* Acute liver disease
* Chronic liver disease unless considered stable for > 6 months.
* Presence of cirrhosis (Child-Pugh Class A, B, or C) or Gilbert's Syndrome.
* Participants with significantly impaired bone marrow function or significant anemia, leukopenia, neutropenia or thrombocytopenia.
* Any concomitant disease that may require chronic treatment with systemic corticosteroids or immunosuppressants during the course of the study.
* History of alcohol or other drug abuse within 12 months prior to screening.
* History of or currently active primary or secondary (non-drug-related) immunodeficiency, including known history of human immunodeficiency virus (HIV) infection.
* Inability to complete an MRI scan.
* Adrenocorticotropic hormone or systemic corticosteroid therapy within 4 weeks prior to screening (inhaled and topical corticosteroids are allowed).
* Receipt of a live-attenuated vaccine within 6 weeks prior to randomization.
* Any previous treatment with immunomodulatory or immunosuppressive medication without an appropriate washout period.

OLE Exclusion Criteria:

* Acute liver disease
* Chronic liver disease unless considered stable for > 6 months

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 746 (Actual)
Dates: Start 2021-03-17 (Actual); Primary Completion 2026-01-27 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Annualized Relapse Rate (ARR) | Minimum of 96 weeks

SECONDARY OUTCOMES:
Time to Onset of Composite 12-week Confirmed Disability Progression (cCDP12) | Minimum of 96 weeks
Time to Onset of Composite 24-week Confirmed Disability Progression (cCDP24) | Minimum of 96 weeks
Time to Onset of 12-week Confirmed Disability Progression (CDP12) | Minimum of 96 weeks
Time to Onset of 24-week Confirmed Disability Progression (CDP24) | Minimum of 96 weeks
Total Number of T1 Gadolinium Enhancing (Gd+) Lesions, New and/or Enlarging T2-weighted Lesions as Detected by Magnetic Resonance Imaging (MRI) | Baseline, Weeks 12, 24, 48 and 96
Percentage Change in Total Brain Volume from Week 24 as Assessed by MRI | From Week 24 to Week 96
Change in Participant-Reported Physical Impacts of Multiple Sclerosis (MS) Measured by the Multiple Sclerosis, 29-Item [MSIS-29] Physical Scale | Baseline, Weeks 12, 24, 36, 48, 60, 72, 84 and 96
  The MSIS-29, Version 2 is a 29-item patient-reported measure of the physical and psychological impacts of MS. Participants are asked to rate how much their functioning and well-being has been impacted over the past 14 days on a 4-point scale, from "Not at all" (1) to "Extremely" (4). The physical score is the sum of items 1-20, which is then transformed to a 0-100 scale. The psychological score is the sum of items 21-29, transformed to a 0-100 scale. Higher scores indicate a greater impact of MS.
Time to Onset of 12-week Confirmed 4-point worsening in Symbol Digit Modality Test (SDMT) Score | Minimum of 96 weeks
  The SDMT is used for detecting the presence of cognitive impairment and changes in cognitive functioning over time and in response to treatment. The SDMT is brief, is easy to administer test, and involves a simple substitution task. Using a reference key, the examinee has 90 seconds to pair specific numbers with given geometric figures. Responses will be collected only orally, and administration time is approximately 5 minutes. The number of correct responses in 90 seconds will be considered the SDMT score. A decrease by 4 points on the SDMT score from baseline represents a clinically meaningful change in cognitive processing. The SDMT score ranges from 0 to 110. The higher the results, the better processing speed/working memory.
Change from Baseline to Week 48 in the Concentration of Blood Neurofilament Light Chain (NfL) | Up to 48 weeks
Percentage of Participants with Adverse Events (AEs) | Up to 4.5 years
Plasma Concentrations of Fenebrutinib at Specified Timepoints | Up to 4.5 years
Time to Onset of Composite 12-week Confirmed Progression Independent of Relapse Activity (cPIRA12) | Minimum of 96 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (160):
- United States (32):
  - University of Alabama Birmingham, Birmingham, Alabama
  - Alabama Neurology Associates, Homewood, Alabama
  - Center for Neurology and Spine - Phoenix - Hunt - PPDS, Phoenix, Arizona
  - Profound Research, LLC, Carlsbad, California
  - University of California Irvine, Irvine, California
  - SC3 Research Group, Inc, Pasadena, California
  - University of Colorado Denver, Aurora, Colorado
  - Mountain View Clinical Research, Denver, Colorado
  - Advanced Neurology of Colorado, LLC, Fort Collins, Colorado
  - Neurology Associates, PA; Research Department, Maitland, Florida
  - NorthShore University HealthSystem, Highland Park, Illinois
  - Fort Wayne Neurological Center, Fort Wayne, Indiana
  - The NeuroMedical Center, Baton Rouge, Louisiana
  - Ochsner LSU Health, Shreveport, Louisiana
  - Johns Hopkins University School Of Medicine; Outpatient Center, Baltimore, Maryland
  - University of Massachusetts Medical School, Worcester, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - Holy Name Hospital; Institute For Clinical Research, Teaneck, New Jersey
  - University of New Mexico; MS Specialty Clinic, Albuquerque, New Mexico
  - Miami Valley Hospital South; Dayton Physician's Office, Centerville, Ohio
  - OhioHealth, Columbus, Ohio
  - The Boster Center for Multiple Sclerosis a Singlepoint Healthcare Company, Columbus, Ohio
  - Oklahoma Medical Research Foundation; MS Center of Excellence, Oklahoma City, Oklahoma
  - St. Luke's University Health network, Bethlehem, Pennsylvania
  - Premier Neurology, Greenville, South Carolina
  - New Orleans Center for Clinical Research, Knoxville, Tennessee
  - North Texas Institute of Neurology and Headache NextStage Clinical Research Clinic, Plano, Texas
  - Texas Institute for Neurological Disorders, Sherman, Texas
  - Multiple Sclerosis Center of Greater Washington, Vienna, Virginia
  - Evergreen MS Center, Kirkland, Washington
  - Wheaton Franciscan Healthcare - St. Francis Outpatient Center; Center for Neurological Disorders, Milwaukee, Wisconsin
- Argentina (7):
  - Instituto de Investigaciones Metabolicas (Idim), Buenos Aires
  - IME - Instituto Médico Especializado, Buenos Aires
  - Centro de Especialidades Neurológicas y Rehabilitación - CENyR, Buenos Aires
  - CIER, C. A. B. A.
  - Diagnostico Medico Oroño, Rosario
  - Cer San Juan, San Juan
  - Centro de Investigaciones Médicas Tucuman, San Miguel de Tucumán
- China (17):
  - Peking University First Hospital, Beijing
  - Beijing Tiantan Hospital,Capital Medical University, Beijing
  - the First Hospital of Jilin University, Changchun
  - Xiangya Hospital Central South University, Changsha
  - West China Hospital, Sichuan University, Chengdu
  - The First Affiliated Hospital, Chongqing Medical University, Chongqing
  - The First Affiliated Hospital of Sun Yat-sen University, Guangzhou
  - The second Affiliated Hospital of Guangzhou Medical University, Guangzhou
  - The affiliated Hospital of Guiyang Medical College, Guiyang
  - The First People?s Hospital of Yunnan Province, Kunming
  - The Second Hospital of Hebei Medical University, Shijiazhuang
  - The First Affiliated Hospital of Soochow University, Suzhou
  - 1st Affiliated Hospital of Shanxi Medical University, Taiyuan
  - Tianjin Medical University General Hospital, Tianjin
  - Xinjiang People Hospital, Ürümqi
  - Tongji Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan
  - Tangdu Hospital, The Fourth Military Medical University, Xi'an
- Dominican Republic (2):
  - NeuroINC, Santiago de los Caballeros
  - Hospital Padre Billini, Santo Domingo
- Helsinki University Central Hospital, Helsinki, Finland
- Georgia (5):
  - New Hospitals, Tbilisi
  - Pineo Medical Ecosystem, Tbilisi
  - St. Michael hospital, Tbilisi
  - MediClab Georgia, Tbilisi
  - Khechinashvili University Hospital, Tbilisi
- Germany (9):
  - Jüdisches Krankenhaus Berlin, Berlin
  - Studienzentrum Dr. Bischof GmbH, Böblingen
  - Universitätsklinikum "Carl Gustav Carus", Zentrum für Klinische Neurowissenschaften, Dresden
  - Universitätsklinikum Gießen und Marburg GmbH, Giessen
  - Uniklinik Schleswig-Holstein, Kiel
  - Praxis Dr. med. Andreas Kowalik, Arzt für Neurologie und Psychiatrie, Stuttgart
  - Universitätsklinikum Tübingen, Zentrum für Neurologie, Tübingen
  - Universitätsklinikum Ulm, Ulm
  - Studienzentrum Nordwest Dr med Joachim Springub Herr Wolfgang Schwarz, Westerstede
- Hong Kong (2):
  - Pamela Youde Nethersole Eastern Hospital, Hong Kong
  - Prince of Wales Hospital, Shatin, New Territories
- Hungary (5):
  - Clinexpert Kft., Budapest
  - S-Medicon Egeszsegugyi Szolgaltato Kft., Budapest
  - Markhot Ferenc Oktatokorhaz és Rendelointezet, Eger
  - Pest Megyei Flor Ferenc Korhaz, Kistarcsa
  - Szegedi Tudományegyetem Szent-Györgyi Albert Klinikai Központ, Szeged
- Italy (12):
  - AO.U. Policlinico Riuniti Foggia, Foggia, Apulia
  - AOU Seconda Università degli Studi, Napoli, Campania
  - AOU Policlinico - Università L. Vanvitelli, Napoli, Campania
  - A.O.U. di Parma, Parma, Emilia-Romagna
  - Policlinico Tor Vergata Dip. Neuroscienze-Clinica Neurologica-UOSD Sclerosi Multipla, Rome, Lazio
  - Policlinico Umberto I, Rome, Lazio
  - Azienda Ospedaliera Sant'Andrea, Rome, Lazio
  - ASST PAPA GIOVANNI XXIII Neurologia USS Malattie Autoimmuni Centro Sclerosi Multipla, Bergamo, Lombardy
  - IRCCS Ospedale San Raffaele, Milan, Lombardy
  - Ospedale Regina Montis Regalis, Mondovì (CN), Piedmont
  - AOU Policlinico V. Emanuele - P.O G. Rodolico, Catania, Sicily
  - Azienda Ospedaliera di Padova, Padua, Veneto
- The Aga Khan University-Kenya., Nairobi, Kenya
- Mexico (5):
  - Clinical Research Institute Saltillo, Saltillo, Coahuila
  - Grupo Medico de Investigacion Clinica Multidisciplinaria, Mexico City, Mexico CITY (federal District)
  - Health Pharma Professional Research, Mexico City, Mexico CITY (federal District)
  - Neurociencias Estudios Clinicos S.C., Culiacán, Sinaloa
  - Hospital General de Mexico, Mexico, Tlaxcala
- Zuyderland Medisch Centrum - Sittard Geleen, Sittard-Geleen, Netherlands
- North Macedonia (3):
  - Clinical Hospital Stip, Shtip
  - PHO General City Hospital 8th September Center for dialysis, Skopje
  - University Clinic for Neurology - Skopje, Skopje
- Peru (6):
  - Hospital IV Alberto Sabogal Sologuren, Bellavista
  - Hospital Nacional Guillermo Almenara Irigoyen, La Victoria, Lima
  - Hospital Nacional Dos de Mayo, Lima
  - Clinica Internacional Sede Lima, Lima
  - Hospital Maria Auxiliadora, Lima
  - Clinica Centenario Peruano Japonesa, Pueblo Libre
- Poland (10):
  - ProNeuro Centrum Medyczne, ?ory
  - Neurocentrum Bydgoszcz sp. z o.o, Bydgoszcz
  - Care Clinic, Katowice
  - MT Medic Krosno, Krosno
  - Centrum Neurologii Krzysztof Selmaj, Lodz
  - Rodzinne Centrum Medyczne Lubimed.pl, Lublin
  - Neurologiczny Niepubliczny ZOZ Centrum Leczenia SM Osrodek Bada? Klinicznych, Plewiska
  - MedPolonia, Poznan
  - Instytut Psychiatrii i Neurologii II Klinika Neurologiczna, Warsaw
  - IBISMED Wielospecjalistyczne Centrum Medyczne, Zabrze
- Portugal (7):
  - Hospital de Braga, Braga
  - HUC, Coimbra
  - Hospital Santo Antonio dos Capuchos, Lisbon
  - Hospital da Luz, Lisbon
  - Hospital Geral de Santo Antonio, Porto
  - Hospital de Sao Joao, Porto
  - Centro Hospitalar Entre o Douro e Vouga E.P.E. - Hospital de São Sebastião, Santa Maria da Feira
- Russia (6):
  - Republican clinical hospital named after G.G. Kuvatov, Ufa, Bashkortostan Republic
  - Leningrad Regional Clinical Hospital, Saint Petersburg, Sankt-Peterburg
  - Pavlov State Medical Uni, Saint Petersburg, Sankt-Peterburg
  - Ulyanovsk Regional Clinical Hospital, Ulyanovsk, Ulyanovsk Oblast
  - Center of Cardiology and Neurology, Kirov
  - FSBIH Siberian Regional Medical Centre of FMBA of Russia, Novosibirsk
- University Clinical Center of Serbia, Belgrade, Serbia
- Spain (11):
  - Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital Quiron de Madrid, Pozuelo de Alarcón, Madrid
  - Hospital Universitario Virgen de Arrixaca, EL Palmar (EL Palmar), Murcia
  - Hospital Alvaro Cunqueiro, Vigo, Pontevedra
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitario de la Princesa, Madrid
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Ramon y Cajal, Madrid
  - Fundacion Jimenez Diaz, Madrid
  - Hospital Regional Universitario de Malaga ? Hospital General, Málaga
  - Hospital Universitario Virgen Macarena, Seville
- Switzerland (2):
  - Inselspital Bern Medizin Neurologie, Bern
  - Ospedale Regionale di Lugano - Civico, Lugano
- Tunisia (3):
  - Hopital Razi, Mannouba
  - Fattouma Bourguiba Hospital, Monastir
  - Hospital Habib Bourguiba, Sfax
- Ukraine (12):
  - MNE Lviv Territorial Medical Association Clinical Hospital for Palliative Care, Lviv, Chernihiv Governorate
  - Salutem Medical Center, Vinnytsia, KIEV Governorate
  - Separated structural unit ?University hospital? of Dnipro State Medical University, Dnipro, Tavria Okruha
  - SI USSRI of Medical and Social Problems of Disabilities of MOHU, Dnipro
  - Ams of Ukraine, Kharkiv
  - Medical Center Dopomoga Plus, Kyiv
  - Medical Center of Private Execution First Private Clinic, Kyiv
  - Lviv Regional Clinical Hospital, Lviv
  - Odesa Regional Clinical Hospital, Odesa
  - Medical Clinical Research Center of Medical Center LLC Health Clinic, Vinnytsi
  - LCC "Medical center "Unimed", Zaporizhzhia
  - Municipal Non-profit Enterprise Zaporizhzhya Regional Hospital Zaporizhzhya Regional Council, Zaporizhzhia

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing